CLINICAL TRIAL: NCT02933710
Title: Postmarketing Surveillance Study for a Live Attenuated Japanese Encephalitis Chimeric Virus Vaccine (IMOJEV®) in Republic of Korea
Brief Title: Postmarketing Surveillance Study for IMOJEV® in Republic of Korea
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: JEC18; U1111-1174-4824 (Other: WHO)
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Japanese Encephalitis
Keywords: Japanese encephalitis; IMOJEV®; Japanese encephalitis chimeric virus vaccine
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- IMOJEV® Vaccine Group: Participants who are 12 months and older and who are given a first dose of IMOJEV® during a routine health care visit

SUMMARY:
The purpose of the study is to perform the re-examination of IMOJEV® in routine clinical settings in accordance with the Ministry of Food and Drug Safety regulation.

Primary objective:

* To describe the safety profile of the first dose of IMOJEV® administered under routine health care visit as primary vaccination or as booster.

DETAILED DESCRIPTION:
Subjects aged 12 months of age and older and who are given study vaccine during routine health-care visits will be enrolled in the study.

No study vaccine will be supplied or administered as part of this study, subjects will be monitored following routine vaccine administration in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed by the subject (for subjects 19 years old and above) or the parent(s) or other legal representative (for subjects under 19 years of age)
* Receipt of the first dose of IMOJEV® (on the day of inclusion) according to approved local insert paper.

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or a medical procedure.
* Subjects who already participated in this study.

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who receive IMOJEV® (either primary or booster dose) during a routine health-care visit
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting solicited injection-site reactions, solicited systemic reactions, unsolicited adverse events, and serious adverse events occurring during the trial | Day 0 up to Day 42 post-vaccination
  Solicited injection-site reactions: Tenderness/Pain, Erythema, and Swelling. Solicited systemic reactions: infants and toddlers (12 to 23 months) Fever (temperature), Vomiting, Abnormal crying, Drowsiness, Loss of appetite and Irritability; Subjects aged 2 years and above, Fever (Temperature), Headache, Malaise, and Myalgia

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- 001, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kim HS, Oh Y, Korejwo J, Castells VB, Yang K. Post-Marketing Surveillance of Adverse Events Following Vaccination with the Live-Attenuated Japanese Encephalitis Chimeric Virus Vaccine (Imojev(R)) in South Korea, 2015-2019. Infect Dis Ther. 2020 Sep;9(3):589-598. doi: 10.1007/s40121-020-00305-6. Epub 2020 May 30. PMID 32474892
- See also: Related Info — http://www.sanofipasteur.com